CLINICAL TRIAL: NCT02308709
Title: Novel Lung Functional Imaging for Personalized Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Tokihiro Yamamoto, Ph.D, Principal Investigator, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 472677; CCRO030 (Other: UC Davis)
Record Dates: First submitted 2014-11-03; First posted 2014-12-04 (Estimated); Results first posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Lung Cancer
Keywords: Radiotherapy; Pulmonary Functional Imaging; Computed Tomography (CT); Image Registration; Functional Image-guided Radiotherapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ventilation image-guided radiotherapy (Experimental): Patients will receive 4D CT ventilation image-guided personalized radiotherapy treatment that selectively avoids irradiating highly-functional lung regions
  Interventions: Radiation: Ventilation image-guided radiotherapy

INTERVENTIONS:
Radiation: Ventilation image-guided radiotherapy — Patient's treatment plan will be created and optimized to minimize the dose to highly-functional lung regions

SUMMARY:
The primary objective of this study is to assess the safety and feasibility of personalized radiotherapy with four-dimensional (4D) computed tomography (CT)-based pulmonary ventilation imaging, which selectively avoids irradiating highly-functional lung regions.

DETAILED DESCRIPTION:
In this clinical trial, the investigators will assess the safety and feasibility of 4D CT ventilation image-guided personalized radiotherapy. The investigators will deliver personalized radiotherapy treatments that selectively avoid irradiating highly-functional lung regions for lung cancer patients, and follow up patients to assess the safety and feasibility. The primary hypothesis to be tested is: 4D CT ventilation image-guided personalized radiotherapy can be delivered safely for lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Primary lung cancer or metastatic disease to the lungs to be treated with either conventionally-fractionated radiotherapy (CFRT) or hypo-fractionated stereotactic ablative radiotherapy (SABR).
* Age restriction and/or gender/ethnic restrictions: Patients must be ≥18 years of age. There are no gender or ethnic restrictions.
* Concurrent chemotherapy is allowed, but not required.
* Life expectancy with treatment should be ≥6 months in the estimation of the treating physicians.
* Zubrod performance status ≤2
* Adequate marrow and hepatic function defined as Hgb ≥8; platelets ≥100k; ANC≥1500; LFTs ≤2x upper limit of normal and creatinine ≤1.3 or creatinine clearance of ≥50
* Patient must be able to provide study specific informed consent prior to study entry.

Exclusion Criteria:

* Prior radiotherapy for thoracic cancer or other malignancy leading to any overlap of planned radiotherapy fields.
* For patients undergoing definitive CFRT, patients with distant metastatic disease are not eligible.
* For patients undergoing SABR, both early stage primary lung cancer patients and those with limited metastatic disease to the lungs are eligible; however, patients with oligometastatic disease should have a controlled primary and no more than one other involved organ system.
* Children (<18 years of age), pregnant women, University of California employees or students, or prisoners will be excluded from this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tokihiro Yamamoto, Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ventilation Image-guided CFRT or SBRT: Patients will receive 4D CT ventilation image-guided personalized radiotherapy treatment that selectively avoids irradiating highly-functional lung regions
  Ventilation image-guided radiotherapy: Patient's treatment plan will be created and optimized to minimize the dose to highly-functional lung regions
Period: Overall Study
Arm/Group | Ventilation Image-guided CFRT or SBRT
Started | 34
Completed | 33
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ventilation Image-guided Radiotherapy
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Grade ≥3 AEs Defined as Definitely, Probably, or Possibly Related to 4D CT Ventilation Image-guided Personalized Radiotherapy
Description: Number of subjects experiencing Grade ≥3 AEs, i.e., Grade ≥3 radiation pneumonitis, grade ≥3 esophagitis, or other grade ≥3 AEs, defined as definitely, probably, or possibly related to 4D CT ventilation image-guided personalized radiotherapy.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Ventilation Image-guided Radiotherapy
Number analyzed (Participants) | 33
participants | 5

2. Secondary Outcome: Radiation Pneumonitis Graded by CTCAE v4.0
Description: Number of participants with Grade ≥ 2 radiation pneumonitis adverse event graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Ventilation Image-guided Radiotherapy
Number analyzed (Participants) | 33
participants | 5

3. Secondary Outcome: Post-treatment Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: The median absolute change from baseline in FEV1 (% predicted) at 6 months after treatment.
Time Frame: Baseline and 6 months
Population: The number of participants analyzed are smaller than 33 due to missing data (disease progression or patient refusal was the main reason).
Measure: Median (Full Range); unit: Percent of predicted FEV1
Groups:
- Ventilation Image-guided SBRT: Patients who receive 4D CT ventilation image-guided personalized radiotherapy treatment that selectively avoids irradiating highly-functional lung regions and who receive stereotactic body radiotherapy (SBRT).
  Ventilation image-guided radiotherapy: Patient's treatment plan will be created and optimized to minimize the dose to highly-functional lung regions
- Ventilation Image-guided CFRT: Patients who receive 4D CT ventilation image-guided personalized radiotherapy treatment that selectively avoids irradiating highly-functional lung regions and who receive conventionally fractionated radiotherapy (CFRT).
  Ventilation image-guided radiotherapy: Patient's treatment plan will be created and optimized to minimize the dose to highly-functional lung regions
Arm/Group | Ventilation Image-guided SBRT | Ventilation Image-guided CFRT
Number analyzed (Participants) | 8 | 11
Percent of predicted FEV1 | 6 [-2 to 23] | -1 [-16 to 10]

4. Secondary Outcome: Post-treatment Change in Diffusing Capacity of the Lung for Carbon Monoxide (DLCO)
Description: The median absolute change from baseline in DLCO (% predicted) at 6 months after treatment.
Time Frame: Baseline and 6 months
Population: as for outcome 3
Measure: Median (Full Range); unit: Percent of predicted DLCO
Arm/Group | Ventilation Image-guided CFRT | Ventilation Image-guided SBRT
Number analyzed (Participants) | 3 | 4
Percent of predicted DLCO | -10 [-27 to 6] | -0.5 [-4 to 9]

ADVERSE EVENTS:
Time Frame: Serious and other adverse events assessed for up to 12 months after treatment is completed, an average of 2 years. All cause mortality assessed for up to about 2.5 year after treatment complete.
Arm/Group | Ventilation Image-guided Radiotherapy
All-Cause Mortality (participants affected / at risk) | 22/33
Serious Adverse Events (participants affected / at risk) | 2/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ventilation Image-guided Radiotherapy (N=33)
Esophagitis (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ventilation Image-guided Radiotherapy (N=33)
Anemia (Blood and lymphatic system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Blurred vision (Eye disorders) | 2
Chest pain (Cardiac disorders) | 3
Chest wall pain (Cardiac disorders) | 3
Constipation (Gastrointestinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 18
Creatinine increased (Investigations) | 4
Dehydration (Metabolism and nutrition disorders) | 5
Depression (Psychiatric disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 7
Dermatitis radiation (Injury, poisoning and procedural complications) | 3
Diarrhea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16
Edema limbs (General disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Esophagitis (Gastrointestinal disorders) | 17
Fatigue (General disorders) | 24
Fever (General disorders) | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Globus sensation (Respiratory, thoracic and mediastinal disorders) | 3
Headache (Nervous system disorders) | 3
Hematuria (Renal and urinary disorders) | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Insomnia (Psychiatric disorders) | 4
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 3
Lymphocyte count decreased (Investigations) | 4
Nausea (Gastrointestinal disorders) | 8
Neutrophil count decreased (Investigations) | 2
Non-cardiac chest pain (General disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5
Pneumonitis (radiographic) (Respiratory, thoracic and mediastinal disorders) | 6
Proteinuria (Renal and urinary disorders) | 2
Pulmonary fibrosis (radiographic) (Respiratory, thoracic and mediastinal disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4
White blood cell decreased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT02308709/Prot_SAP_000.pdf